CLINICAL TRIAL: NCT03072615
Title: Role of SWE-change After TIPS in the Prediction of Prognosis After TIPS
Acronym: TIPS-SWE
Status: Completed | Type: Observational
Sponsor: Jonel Trebicka (Other)
Responsible Party: Sponsor-Investigator, Jonel Trebicka, Prof. Dr., University Hospital, Bonn
Organization: University Hospital, Bonn (Other)
Other Study IDs: TIPS-SWE
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Portal Hypertension; Liver Cirrhoses
MeSH Terms: conditions — Hypertension, Portal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: receiving TE before and 30 min after TIPS
  Interventions: Diagnostic Test: Stiffness measurement
- 2: receiving SWE before and 7 days, 6 weeks and 3 months after TIPS
  Interventions: Diagnostic Test: Stiffness measurement

INTERVENTIONS:
Diagnostic Test: Stiffness measurement — Transient Elastopgraphy (TE) or Shear-Wave-Elastography

SUMMARY:
The aim of our prospective multicenter study was to investigate the prognostic value of the acute and long-term changes of liver stiffness in patients receiving a transjugular intrahepatic portosystemic shunt (TIPS).

DETAILED DESCRIPTION:
We included 83 patients receiving TIPS for prevention of rebleeding, therapy-refractory ascites or both. Hemodynamic parameters were assessed before TIPS and after TIPS insertion. 16 patients from Freiburg underwent TE immediately before and after TIPS. In 67 patients from Bonn, SWE of liver and spleen, as well as clinical and biochemical parameters were assessed before TIPS, seven days and six weeks after TIPS.

ELIGIBILITY:
Inclusion Criteria:

* TIPS insertion and had reliable SWE or TE measurement

Exclusion Criteria:

* contraindication for TIPS
* no reliable SWE or TE measurement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This prospective multicentre study included patients, which underwent TIPS insertion and had reliable SWE or TE measurement of the liver before TIPS.
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2013-04-01 (Actual); Primary Completion 2015-11-30 (Actual); Study Completion 2016-02-29 (Actual)

PRIMARY OUTCOMES:
Survival | 3 months

SECONDARY OUTCOMES:
Acute-on-chronic Lvier failure | 3 months

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jansen C, Moller P, Meyer C, Kolbe CC, Bogs C, Pohlmann A, Schierwagen R, Praktiknjo M, Abdullah Z, Lehmann J, Thomas D, Strassburg CP, Latz E, Mueller S, Rossle M, Trebicka J. Increase in liver stiffness after transjugular intrahepatic portosystemic shunt is associated with inflammation and predicts mortality. Hepatology. 2018 Apr;67(4):1472-1484. doi: 10.1002/hep.29612. Epub 2018 Feb 20. PMID 29059466